CLINICAL TRIAL: NCT04993612
Title: Blood Gas Analysis Obtained in Pulmonary Capillary Wedge Position During Right Heart Catheterization
Brief Title: Postcapillary Blood Gas Analysis in Wedge Position (Wedge-BGA)
Status: Recruiting | Type: Observational
Sponsor: Ayham Daher (Other)
Responsible Party: Sponsor-Investigator, Ayham Daher, Principal Investigator, RWTH Aachen University
Organization: RWTH Aachen University (Other)
Other Study IDs: 21-063
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- No pulmonary Hypertension
  Interventions: Diagnostic Test: Blood gas analysis
- pulmonary Hypertension Group 1
  Interventions: Diagnostic Test: Blood gas analysis
- pulmonary Hypertension Group 2
  Interventions: Diagnostic Test: Blood gas analysis
- pulmonary Hypertension Group 3
  Interventions: Diagnostic Test: Blood gas analysis
- pulmonary Hypertension Group 4
  Interventions: Diagnostic Test: Blood gas analysis
- pulmonary Hypertension Group 5
  Interventions: Diagnostic Test: Blood gas analysis

INTERVENTIONS:
Diagnostic Test: Blood gas analysis — Two blood samples will be drawn from the "wedge" position", behind the inflated balloon, during the right heart catheterization, and blood gas analyses will be performed. First sample will be drawn directly after inflating the ballon, and the second one 2 minutes later.

SUMMARY:
If pulmonary hypertension is suspected, a right heart catheterization is usually performed to confirm or rule out the diagnosis. As part of this examination, blood samples are taken from various locations as standard and blood gas analyses are performed. One of the most important measurements during the right heart catheterization is the measurement of the pulmonary arterial occlusion pressure by the so-called wedge maneuver. To measure this value, the catheter with inflated balloon must be advanced into the pulmonary vessels until the "wedge" position is reached, i.e. the balloon completely occludes a branch of the pulmonary artery. In this study, the investigators want to characterize patients with pulmonary hypertension of different causes in more detail. To do that, two blood samples (totaling approximately 4 mL of blood, one sample directly after occlusion and the other one two minutes later) will be drawn during the right heart catheterization from the above-mentioned "wedge" position", behind the inflated balloon, and blood gas analyses will be performed on these samples. In addition, various clinical parameters (comorbidities, etc.) will be recorded by means of clinical questionnaires. Follow-up data will be analyzed and correlations with the aforementioned blood gas analyses will be examined. The results of the study will be used to more precisely characterize the still vague concept of secondary pulmonary hypertension. This could help to develop new therapeutic strategies in some subgroups in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a clearly defined indication for Right heart catheterization.
* Age > 18 years
* Informed consent for participation in the study will sign

Exclusion Criteria:

* Individuals who are not fully capable of giving consent and understanding the nature, significance, and scope of the study
* Pregnancy and lactation
* Wedge-BGA not possible

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving right heart catheterization for appropriate indications will be interviewed for their consent to participate in the study
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Between group differences | At the time of recruitment
  Differences in the Wedge-BGA between groups

SECONDARY OUTCOMES:
Follow-up | 1 and 5 years
  Risk stratification and mortality after 1 and 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital RWTH Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Undecided